CLINICAL TRIAL: NCT07021092
Title: PERSON-CENTERED APPROACHES TO VIREMIA: CONNECTION, RAPPORT, AND ENGAGEMENT STUDY
Acronym: P-CoRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIDRZ; INV-050580 (Other Grant/Funding Number: Gate Foundation)
Record Dates: First submitted 2025-03-25; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HIV Viremia; HIV -1 Infection
Keywords: Uncontrolled Viremia; Person Centred Care; Unmonitored Viral Load
MeSH Terms: interventions — Association

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracing to Ascertain Outcome (Other)
  Interventions: Other: Interventions will be developed in aim 2 of the study.

INTERVENTIONS:
Other: Interventions will be developed in aim 2 of the study. — Person-centred package that connects patients to service delivery, builds rapports and improves engagement in care leading to sustained viral load suppressions
  Other Names: Possible interventions to be developed will include 1) community- based outreach and in-person tracing to identify and establish contact with viremic patients and establish barriers to care; Improved counselling using PCC and being non-judgemental as a way of establishing rapport and relationship with individuals using PCC approach tailored to barriers; Facility based Viral load champions, couple counselling and access to DSD models as a way of providing structural interventions to bring individuals back to care, keep them in care and maintain VL sup

SUMMARY:
The study aims to increase the reach of the person-centred interpersonal practices by developing and accessing a tailored, scalable, and sustainable approach that meets the distinctive needs of populations identified as most disproportionately affected by viremia in Zambia. The study population include pregnant and breastfeeding women, children, adolescents and adult that are more than thirty -30 days late for their next hospital appointments.The study will be implemented over a period of 36 months in 24 facilities in Lusaka and Central province, Zambia.

DETAILED DESCRIPTION:
The study has three aims, that include (1) To assess barriers to sustained viral suppression through identifying prevailing pathways to viremia (2) Apply Human Centred Design methods with stakeholders to co-create person-centred pathways to strengthen viral suppression, with particular attention to vulnerable groups (3) To test P-CoRE package with a focus on high- priority populations contributing to remaining viremia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that are lost to follow up ([LTFU] from HIV care i.e. confirmed >30 days late for a scheduled appointment) at the time of sampling. (i.e. not people who were previously LTFU but then returned and have a documented VL.)
2. Individuals returning to care after being out of care and not taking ART with no VL measure (i.e., unmeasured viremia)
3. Patients that are 6 months late for a scheduled Viral Load (VL) according to Ministry of Health guidelines at the time of sampling (regardless of care status)
4. Patients that have a last documented VL that is elevated, > 1000 copies/ml at time of sampling in current clinic population (CCP) (regardless of care status)
5. Participant that are willing to provide written informed consent in English, or any of the local languages that include Nyanja or Bemba.

Exclusion Criteria:

1. Patients that are unable to provide consent or unwilling to participate in the study
2. Participant who is NOT living with HIV/AIDS;
3. Participant is too sick i.e., failing to talk, general discomfort and emergency cases);

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Updated Estimates of Viremia and Care Status | 2 years
  The study will use a sampling based approach for outcome ascertainment as used in the Better Information for Health in Zambia(BetterInfo) study https://www.cidrz.org/wp-content/toolkits/betterinfo/, but adapt procedures so they are focused on assessments of viremia (rather than mortality as in the initial BetterInfo study) (21). This approach leverages data collected during routine care and augments it with targeted data collection in a smaller sample of clients with incomplete data (i.e., missing VL measurements) to provide robust and epidemiologically rigorous estimates for the full clinic population.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aaloke Mody, Principal Investigator — Washington University School of Medicine; Kombatende Sikombe, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (2):
- Zambia (2):
  - Ministry of Health, Lusaka, Lusaka Province
  - Railway GRZ Urban Health Centre, Kafue District Health Hospital, Nangongwe OPD Urban Health Centre, Chawama 1st level hospital, Chipate 1st level hospital, Matero Reference Health Centre, Mtendere Health Centre, Lwiimba Rural Health Centre, Lusaka, Lusaka Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrenkranz P, Rosen S, Boulle A, Eaton JW, Ford N, Fox MP, Grimsrud A, Rice BD, Sikazwe I, Holmes CB. The revolving door of HIV care: Revising the service delivery cascade to achieve the UNAIDS 95-95-95 goals. PLoS Med. 2021 May 24;18(5):e1003651. doi: 10.1371/journal.pmed.1003651. eCollection 2021 May. PMID 34029346
- See also: The study will use similar procedures for a sampling based approach for outcome ascertainment as that used in the Better Information for Health in Zambia Study. — https://www.cidrz.org/wp-content/toolkits/betterinfo/
- See also: Related Info — https://www.cidrz.org/wp-content/toolkits/betterinfo/